CLINICAL TRIAL: NCT03006458
Title: A Clinical Comparison of the Comfilcon A (Extended Range) XR Toric Multifocal and Omafilcon B Toric XR Multifocal Contact Lenses
Brief Title: A Clinical Comparison of 2 Multifocal Toric XR (Extended Range) Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CV-16-28 (C16-599)
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Results first posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- comfilcon A (Experimental): Participants were randomized to wear comfilcon A toric lenses for two weeks during the cross over study.
  The final optical design of comfilcon A contact lens was optimized to improve the quality and two further studies (CV-18-10 and CV-18-11) were conducted after completion of this study to evaluate the modified optical design.
  Interventions: Device: comfilcon A
- omafilcon B (Active Comparator): Participants were randomized to wear omafilcon B toric lenses for two weeks during the cross over study.
  Interventions: Device: omafilcon B

INTERVENTIONS:
Device: comfilcon A — toric contact lens
  Arms: comfilcon A
Device: omafilcon B — toric contact lens
  Arms: omafilcon B

SUMMARY:
This study aims to compare the clinical performance and subjective acceptance of the comfilcon A and the omafilcon B soft contact lenses.

DETAILED DESCRIPTION:
This will be a randomized, subject-masked, crossover, bilateral study, controlled by cross comparison. Thirty subjects will use each lens type for two weeks in random sequence. Follow-up visits for each lens will be performed after two weeks of wear. Lenses will be worn on a daily wear basis.

The final optical design of comfilcon A contact lens was optimized to improve the quality and two further studies (CV-18-10 and CV-18-11) were conducted after completion of this study to evaluate the modified optical design.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will only be eligible for the study if:

  1. They are aged 40 - 70 years, inclusive.
  2. They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
  3. They are willing and able to follow the protocol.
  4. They have successfully completed the non-dispensing study (C16-597) as the lenses to be worn on this study (C16-599) are predetermined from their participation on study C16-597.
  5. They have a contact lens spherical prescription between +10.00 to -10.00D (Diopters) (inclusive).
  6. They have astigmatism between of -0.75 and -5.75DC (based on the calculated ocular refraction) in each eye.
  7. They have an Add component to their spectacle refraction (between +0.75 and

     +2.50DS).
  8. They can be satisfactorily fitted with the study lenses.
  9. They can attain at least 0.30 logMAR binocular distance high contrast visual acuity with the study lenses within the available power range.
  10. They have successfully worn soft contact lenses in the last two years.
  11. They are willing to comply with the wear schedule (at least five days per week and for at least six hours per day).
  12. They agree not to participate in other clinical research for the duration of this study.
  13. They own a wearable pair of spectacles.

Exclusion Criteria:

* Subjects will not be eligible to take part in the study if:

  1. They have an ocular disorder which would normally contra-indicate contact lens wear.
  2. They have a systemic disorder which would normally contra-indicate contact lens wear.
  3. They are using any topical medication such as eye drops or ointment.
  4. They have had cataract surgery.
  5. They have had corneal refractive surgery.
  6. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
  7. They are pregnant or breast-feeding.
  8. They have any clinically meaningful slit lamp findings contraindicating contact lens wear (e.g. ≥ Grade 3 finding of oedema, corneal neovascularisation, corneal staining, tarsal abnormalities, conjunctival injection, blepharitis/meibomian gland dysfunction) on the Efron classification scale or any other ocular abnormality that in the opinion of the investigator would contraindicate contact lens wear.
  9. They have any infectious disease (e.g. hepatitis) which would, in the opinion of the investigator, contraindicate contact lens wear or pose a risk to study personnel; or they have any immunosuppressive disease (e.g. HIV).
  10. They have a history of anaphylaxis or severe allergic reaction.
  11. They have taken part in any other contact lens or care solution clinical trial or research, within two weeks prior to starting this study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-12; Primary Completion 2017-04-06 (Actual); Study Completion 2017-04-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eurolens Research, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Comfilcon A Then Omafilcon B: Participants were randomized to wear comfilcon A for two weeks during the cross over study.
  comfilcon A: toric contact lens
- Omafilcon B Then Comfilcon A: Participants were randomized to wear omafilcon B for two weeks during the cross over study.
  omafilcon B: toric contact lens
Period: First Intervention
Arm/Group | Comfilcon A Then Omafilcon B | Omafilcon B Then Comfilcon A
Started | 14 | 10
Completed | 14 | 7
Not Completed | 0 | 3
Not completed — Unsatisfied Vision | 0 | 3
Period: Second Intervention
Arm/Group | Comfilcon A Then Omafilcon B | Omafilcon B Then Comfilcon A
Started | 14 | 10
Completed | 14 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Total Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 24

OUTCOME MEASURES:

1. Primary Outcome: Stability
Description: Investigator's acceptance on overall stability for comfilcon A and omafilcon B lenses assessed using grading scale 0-4, 0=Totally unstable, can't be worn to provide acceptable vision correction for astigmatism, 4=Excellent orientation and optimum rotational.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Comfilcon A: Participants were randomized to wear comfilcon A toric lenses for two weeks during the cross over study.
  comfilcon A: toric contact lens
Arm/Group | Comfilcon A | Omafilcon B
Number analyzed (Participants) | 24 | 21
units on a scale | 3.2 (1.5) | 2.9 (0.9)

2. Primary Outcome: Stability
Description: as for outcome 1
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Omafilcon B
Number analyzed (Participants) | 24 | 21
units on a scale | 3.2 (0.7) | 2.5 (1.0)

3. Primary Outcome: Overall Toric Lens Fit Acceptance
Description: Overall toric lens fit acceptance is assessed for comfilcon A and omafilcon B lenses. Scale 0-4, 0=can't be worn, 1=Poor, 2=Fair, 3=Good, 4=optimum.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Omafilcon B
Number analyzed (Participants) | 24 | 21
units on a scale | 3.3 (0.5) | 3.2 (0.6)

4. Primary Outcome: Overall Toric Lens Fit Acceptance
Description: as for outcome 3
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Omafilcon B
Number analyzed (Participants) | 24 | 21
units on a scale | 3.5 (0.6) | 2.8 (0.7)

5. Primary Outcome: Comfort
Description: Subjective ratings for comfort assessed. Scale 0-100, 0=cannot be worn, causes pain; 100=cannot be felt ever
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Omafilcon B
Number analyzed (Participants) | 24 | 21
units on a scale | 81.6 (20.3) | 79.7 (21.6)

6. Primary Outcome: Comfort
Description: Subjective ratings for comfort assessed. Scale 0-100, 0=cannot be worn, causes pain; 100=cannot be felt ever
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Omafilcon B
Number analyzed (Participants) | 24 | 21
units on a scale | 79.8 (21.8) | 70.6 (27.2)

7. Primary Outcome: Overall Satisfaction
Description: Subjective ratings for overall satisfaction for comfilcon A and omafilcon B lenses assessed. Scale 0-100, 0=extremely dissatisfied, 100=extremely satisfied
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Omafilcon B
Number analyzed (Participants) | 24 | 21
units on a scale | 63.0 (31.4) | 63.3 (34.4)

8. Primary Outcome: Dryness
Description: Subjective ratings for dryness assessed. Scale 0-100, 0=cannot be worn, extremely dry; 100=no dryness experienced at any time
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Omafilcon B
Number analyzed (Participants) | 24 | 21
units on a scale | 80.4 (24.7) | 77.2 (24.1)

9. Primary Outcome: Visual Fluctuation/ Stability
Description: Subjective ratings for visual fluctuation/stability assessed. Scale 0-100, 0=totally unstable/ fluctuation/changing; 100=perfectly stable/not fluctuation/changing
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Omafilcon B
Number analyzed (Participants) | 24 | 21
units on a scale | 81.0 (16.1) | 73.8 (25.5)

10. Primary Outcome: Handling
Description: Subjective ratings for handling difficulty assessed at 2 weeks. Scale 0-100, 0=very difficult, 100=very easy
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Omafilcon B
Number analyzed (Participants) | 24 | 21
units on a scale | 84.5 (15.0) | 85.8 (17.1)

11. Primary Outcome: Quality of Near Vision
Description: Subjective ratings for quality of near vision. Scale 0-100, 0=extremely poor vision all of the time. cannot function, 100 - excellent vision all of the time.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Omafilcon B
Number analyzed (Participants) | 24 | 21
units on a scale | 38.5 (30.5) | 56.4 (28.9)

12. Primary Outcome: Quality of Intermediate Vision
Description: Subjective ratings for quality of intermediate vision. Scale 0-100, 0=extremely poor vision all of the time. cannot function, 100 - excellent vision all of the time.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Omafilcon B
Number analyzed (Participants) | 24 | 21
units on a scale | 50.2 (29.5) | 65.3 (25.6)

13. Primary Outcome: Quality of Distance Vision
Description: Subjective ratings for quality of distance vision. Scale 0-100, 0=extremely poor vision all of the time. cannot function, 100 - excellent vision all of the time.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Omafilcon B
Number analyzed (Participants) | 24 | 21
units on a scale | 86.2 (13.7) | 67.3 (25.5)

14. Primary Outcome: Quality of Vision While Driving During the Day
Description: Subjective rating for quality of vision while driving during the day. Scale 0-100, 0=extremely poor vision all of the time. cannot function, 100 - excellent vision all of the time.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Omafilcon B
Number analyzed (Participants) | 20 | 17
units on a scale | 87.3 (14.6) | 76.2 (25.4)

15. Primary Outcome: Quality of Vision While Driving During the Night
Description: Subjective ratings for quality of vision while driving at night. Scale 0-100, 0=extremely poor vision all of the time. cannot function, 100 - excellent vision all of the time.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Omafilcon B
Number analyzed (Participants) | 20 | 15
units on a scale | 78.0 (18.6) | 67.0 (23.4)

16. Primary Outcome: Ghosting at Near
Description: Subjective ratings for ghosting at near assessed at 2 weeks. Scale 0-100, 0=intolerable, 100=not noticeable.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Omafilcon B
Number analyzed (Participants) | 23 | 21
units on a scale | 66.5 (35.0) | 78.1 (27.0)

17. Primary Outcome: Ghosting at Distance
Description: Subjective ratings for ghosting at distance assessed at 2 weeks. Scale 0-100, 0=intolerable, 100=not noticeable.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Omafilcon B
Number analyzed (Participants) | 24 | 21
units on a scale | 83.3 (24.8) | 86.9 (24.4)

ADVERSE EVENTS:
Time Frame: From baseline to follow up visit for an average of 2 weeks.
Arm/Group | Comfilcon A | Omafilcon B
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 0/24 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/58/NCT03006458/Prot_SAP_000.pdf